CLINICAL TRIAL: NCT02100371
Title: Extension Protocol of BMS-833923 in Subjects With Basal Cell Nevus Syndrome
Brief Title: Study of BMS-833923 in Two Specific Patients With Basal Cell Nevus Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA194-103
Record Dates: First submitted 2014-02-28; First posted 2014-03-31 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Basal Cell Nevus Syndrome
Keywords: BMS-833923; CA194002
MeSH Terms: conditions — Basal Cell Nevus Syndrome | interventions — BMS-833923

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-833923 (Experimental): BMS-833923, by mouth, at the dose and schedule administered while enrolled in CA194002.
  Interventions: Drug: BMS-833923

INTERVENTIONS:
Drug: BMS-833923 — BMS-833923, by mouth, at the dose and schedule administered while enrolled in CA194002.
  Other Names: XL139

SUMMARY:
This is an extension study of Protocol CA194002 to allow 2 specific participants with basal cell nevus syndrome in the CA194002 study at Princess Margaret Cancer Centre who are still benefitting from the study drug BMS-833923 to continue receiving the study drug. This study will continue to evaluate the safety and tolerability of BMS-833923 in these participants.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of BMS-833923 administered on an extension protocol in subjects with basal cell nevus syndrome (BCNS). This is an extension study of Protocol CA194002 to allow 2 specific participants with BCNS in the CA194002 study at Princess Margaret Cancer Centre who are still benefitting from the study drug BMS-833923, to continue receiving the study drug. In this open-label extension protocol, no new subjects will be recruited. The two BCNS subjects from Protocol CA194002 (subjects CA194002-1-14 and CA194002-1-25) will continue to receive BMS-833923 at the dose and schedule administered on CA194002 until fulfilling protocol criteria for discontinuation. These patients are receiving different doses: one being 60mg once every 2 weeks, and the other is receiving 300mg once daily. This study will continue to evaluate the safety and tolerability of BMS-833923 in these participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Two specific study participants enrolled on protocol CA194002 at Princess Margaret Cancer Centre and remain on BMS-833923 at the time of study entry
* Women, age 18 years and above
* Agree to use methods to prevent pregnancy, not pregnant or breastfeeding

Exclusion Criteria:

* Known symptomatic brain metastasis
* A serious uncontrolled medical disorder or active infection, which would impair the ability of the patient to receive protocol therapy
* Gastrointestinal disease or surgery that could impact the absorption of study drug
* Inability to swallow oral medication
* Inability to be venipunctured and/or tolerate venous access
* Uncontrolled or significant cardiovascular
* Any other medical, psychiatric and/or social reason
* Have HIV, HepB, or HepC
* Exposure to immunosuppressants and immunotherapy concurrently with study treatment and up to 3 months
* Acceptable physical and laboratory test findings
* History of allergy to compounds chemically-related

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Frequency of side effects experienced per participant | From date of first study drug dose taken for this study until participant discontinuation, assessed up to 5 years

SECONDARY OUTCOMES:
Length of time participants' disease does not worsen | From date of first study drug dose taken for this study until the date of first documented progression or date of death from any cause, whichever comes first, accessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada